Recovery Management Checkups for Primary Care (RMC-PC) Experiment

NCT 1119-1216

September 7, 2018

## Informed Consent Recovery Management Checkups for Primary Care (RMC-PC) Draft 9/7/18

**Why are you doing this study?** To see if we can help get people with a drug or alcohol problem get into treatment. We also want to see if that helps make their lives better.

What will happen? You will be interviewed 1 to 5 days after your visit at the health center. Other interviews will take place every 3 months for a year. All interviews will take place face to face. You will be asked to give us phone numbers and addresses so we can stay in touch with you. You will be photographed once by project staff, and the photograph will be attached to your Locator Form. The photograph will help project staff verify that the person they are interviewing each time is in fact you and not someone else. This photograph is also used to identify and locate you for follow-up interview purposes, and it may be shown to individuals to help locate you. These individuals will only be told that the researchers are trying to locate you for a health study in which you have agreed to participate. At the end of the project and after all follow-up interviews have been completed, a member of the project team will destroy the photograph.

**What takes place at an interview?** We ask you questions for about 30-45 minutes. You can say no if you do not want to answer any question. You will also be asked to give a urine sample for testing. You will receive a \$35 visa card for each interview and another \$15 visa gift card for the urine test. The total you can get for each interview is a \$50 visa card.

**How is the study organized?** You will be placed into 1 of 2 groups. One group will only do interviews. The other group will do interviews and will receive help getting into treatment. No matter if you are in group 1 or group 2, you can always go to treatment and community-based recovery support services as usual.

How will information about me be shared with others? Your name and other information about you like your date of birth will be taken out of your file before it is given to anyone else. Your information will not be made public in any way. We have a **Certificate of Confidentiality** from the National Institutes of Health. It means we cannot be "forced" to give out any information to anyone that tells them you are in this study. We would only share information about you if you tell us you are going to hurt yourself or others. We also would share your information if you tell us about a time when you hurt an older person or if you hurt or left a child uncared for.

What risks am I taking? There is a chance that some information about you could be found out. This is not usually a problem. Staff people who work on these studies need to follow federal laws. The federal laws protect your information. The people who interview you know how to protect your information. They must follow the rules in the **Certificate of Confidentiality**.

What if I want to quit the study? You may take yourself out of the study at any time. You must give a written note to the person who is in charge of the study. You will still be able to go to your usual treatment or recovery services. When you stay in this study and take part in the interviews, you are helping us understand people with drug and alcohol problems. Your answers to questions are important and give us helpful ideas.

I agree to take part in the study: The study has been explained to me. I had a chance to ask questions. I understand that I can choose not to answer any question and that I can take myself out of this study at any time. I will be can continue with my usual treatment even if am not in the study. No one has made any promises about how the study will turn out. My personal

| information related to the study will be prote<br>When my information is looked at for a requ<br>be protected by federal laws. | | |
|---|---|---|
| I hereby agree / do not agree (che this consent form. I have been given a copy questions or concerns, I can contact the macharge is Dr. Christy Scott (Phone: 312-664 cscott@chestnut.org). If I have questions all can contact the person in charge of protections. | of the consent form. I understand the<br>ain person in charge of the study. The<br>1-4321, Fax: 312-274-5335, e-mail:<br>bout my rights as a person in this rese | at if I have<br>person in<br>earch study, I |
| Participant (please print) | Participant (signature) | Date |
| Witness (signature) | Date | |
| IneligibleRefused (Reason: | ) | |